CLINICAL TRIAL: NCT01983787
Title: Pharmacokinetics of Piperacillin, Given as Continuous Infusion to Patients With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Kristina Öbrink-Hansen, MD, University of Aarhus
Other Study IDs: CF-275-13
Record Dates: First submitted 2013-07-11; First posted 2013-11-14 (Estimated); Results first posted 2015-10-01 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Continuous infusion; Pharmacokinetics
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pharmacokinetics Piperacillin: Patients with cystic fibrosis , treated with Piperacillin/Tazobactam, given as continuous infusion for a period of two weeks.

SUMMARY:
At the Department of Infectious Diseases, Aarhus University Hospital, continuous infusion with piperacillin/tazobactam for a period of 2 weeks, has been used for several years in patients with cystic fibrosis, suffering from acute pulmonary exacerbations (APE).

It is an outpatient treatment. To assess the efficacy and quality of the treatment, a blood test every 3rd day is taken to determine the concentration of Piperacillin in blood-plasma.

DETAILED DESCRIPTION:
Patients with cystic fibrosis (CF) are often colonized with multidrug-resistant microorganisms, which increases the risk of suboptimal dosing of antibiotics as the time above the minimum inhibitory concentration (T>MIC) is suboptimal. Continuous infusion of beta-lactam antibiotics is more likely to optimize T>MIC than intermittent infusion. At the Department of Infectious Diseases, Aarhus University Hospital, continuous infusion with piperacillin/tazobactam for a period of 2 weeks, has been used for several years in patients with CF, suffering from acute pulmonary exacerbations (APE). It is an outpatient treatment, and the patients are given 16 g of piperacillin per 24 hours. To assess the efficacy and quality of the treatment, a blood test every 3rd day will be required to monitor the blood-plasma concentration of piperacillin, as well as C-reactive protein (CRP) and white blood cell count (WBC).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cystic Fibrosis, suffering from acute pulmonary exacerbations, treated with continuous infusion of Piperacillin/Tazobactam for a period of two weeks.

Exclusion Criteria:

* Age under 18

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Cystic Fibrosis, suffering from acute pulmonary exacerbations.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eskild Petersen, Professor, Study Director — Department of Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus, Aarhus N, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Pharmacokinetics Piperacillin: Patients with cystic fibrosis with pulmonary exacerbation, treated with Piperacillin/Tazobactam, given as continuous infusion for a period of two weeks.
Period: Overall Study
Arm/Group | Pharmacokinetics Piperacillin
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pharmacokinetics Piperacillin: Patients with cystic fibrosis and pulmonary exacerbation, treated with Piperacillin/Tazobactam, given as continuous infusion for a period of two weeks.
Arm/Group | Pharmacokinetics Piperacillin
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Blood-plasma Concentration of Piperacillin
Description: The free, non-protein bound fraction of plasma piperacillin for each patient was determined using Ultra High Performance Liquid Chromatography. The concentration was compared to the MIC-value (Minimal Inhibitory Concentration) of the pathogen isolated in a sputum sample collected prior to initiation of antibiotic treatment.
  Infusion pumps with 16 g of piperacillin per 24 hours were initially used and five patients had piperacillin plasma-concentrations monitored during this treatment regimen. However, in three of these patients, the piperacillin plasma concentrations were unexpectedly low and dropped to a level below the MIC. This was found to be due to antibiotic crystallization within the infusion pumps as a result of the antibiotic concentration being too high. Consequently, infusion pumps with 12 g of piperacillin per 24 hours were used in stead. The median piperaillin concentrations reported below are derived from all measurements within the two weeks of treatment.
Time Frame: Piperacillin plasma-concentration was determined 3-5 times for each patient, during the 2 weeks of piperacillin treatment
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Pharmacokinetics Piperacillin 16g/Day: Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 16 g/24 hours, given as continuous infusion for a period of two weeks.
- Pharmacokinetics Piperacillin 12g/Day: Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 12 g/24 hours, given as continuous infusion for a period of two weeks.
Arm/Group | Pharmacokinetics Piperacillin 16g/Day | Pharmacokinetics Piperacillin 12g/Day
Number analyzed (Participants) | 5 | 5
mg/L | 21 [5 to 33.5] | 21 [15 to 42]

2. Secondary Outcome: The Time Above the Minimum Inhibitory Concentration (T>MIC)
Description: The time, expressed in percentage, for which the plasma concentration of Piperacillin lies above the minimum inhibitory concentration for the pathogen,during the treatment. If the piperacillin concentration at all measurements during the treatment period was at a level above the MIC, T>MIC is reported as 100%. MIC for the pathogen in sputum was not reported in patient 5. Therefore,T>MIC for this patient could not be estimated.
  Patient 1-5 were treated with piperacillin 16g/day. Patient 6-10 were treated with piperacillin 12g/day.
Time Frame: Patients will be followed for the duration of treatment, which is approximately 2 weeks.
Measure: Number; unit: % of time above the MIC
Groups:
- T>MIC 16g/Day, Patient 1; T>MIC 16g/Day, Patient 4: Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 16 g/24 hours, given as continuous infusion for a period of two weeks. Pathogen in sputum: Staphylococcus aureus. If the piperacillin concentration at all measurements during the treatment period was at a level above the MIC, T>MIC is reported as 100%.
- T>MIC 16g/Day, Patient 2; T>MIC 16g/Day, Patient 3: Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 16 g/24 hours, given as continuous infusion for a period of two weeks. Pathogen in sputum: Pseudomonas aeruginosa. If the piperacillin concentration at all measurements during the treatment period was at a level above the MIC, T>MIC is reported as 100%.
- T>MIC12g/Day, Patient 6; T>MIC 12g/Day, Patient 7; T>MIC 12g/Day, Patient 8; T>MIC 12g/Day, Patient 10: Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 12 g/24 hours, given as continuous infusion for a period of two weeks.Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 16 g/24 hours, given as continuous infusion for a period of two weeks. Pathogen in sputum: Staphylococcus aureus. If the piperacillin concentration at all measurements during the treatment period was at a level above the MIC, T>MIC is reported as 100%.
- T>MIC 12g/Day, Patient 9: Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 12 g/24 hours, given as continuous infusion for a period of two weeks.Patients with cystic fibrosis , treated with Piperacillin/Tazobactam 16 g/24 hours, given as continuous infusion for a period of two weeks. Pathogen in sputum: Acromobacter. If the piperacillin concentration at all measurements during the treatment period was at a level above the MIC, T>MIC is reported as 100%.
Arm/Group | T>MIC 16g/Day, Patient 1 | T>MIC 16g/Day, Patient 2 | T>MIC 16g/Day, Patient 3 | T>MIC 16g/Day, Patient 4 | T>MIC12g/Day, Patient 6 | T>MIC 12g/Day, Patient 7 | T>MIC 12g/Day, Patient 8 | T>MIC 12g/Day, Patient 9 | T>MIC 12g/Day, Patient 10
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
% of time above the MIC | 100 | 100 | 75 | 75 | 100 | 100 | 100 | 100 | 100

3. Secondary Outcome: MIC of Pathogen Detected in Sputum Sample, Prior to Initiation of Treatment.
Description: MIC to piperacillin/tazobactam was obtained by using E-tests (AB Biodisk, Solna, Sweden) on Mueller-Hinton agar plates incubated at 35 ± 2 degrees Celcius with inoculum, incubation time and atmosphere in accordance to the E-test application guide.
Time Frame: Sputum sample was collected 3 to 7 days before treatment initiation.
Measure: Number; unit: mg/L
Groups:
- Patient 1; Patient 4; Patient 7; Patient 8: MIC (mg/L) of pathogen detected in sputum: 3 mg/L
- Patient 2: MIC (mg/L) of pathogen detected in sputum: 8 mg/L
- Patient 3: MIC (mg/L) of pathogen detected in sputum: 16 mg/L
- Patient 6: MIC (mg/L) of pathogen detected in sputum: 0.5 mg/L
- Patient 9: MIC (mg/L) of pathogen detected in sputum: 0.75 mg/L
- Patient 10: MIC (mg/L) of pathogen detected in sputum: 2 mg/L
Arm/Group | Patient 1 | Patient 2 | Patient 3 | Patient 4 | Patient 6 | Patient 7 | Patient 8 | Patient 9 | Patient 10
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
mg/L | 3 | 8 | 16 | 3 | 0.5 | 3 | 3 | 0.75 | 2

ADVERSE EVENTS:
Arm/Group | Pharmacokinetics Piperacillin
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes